CLINICAL TRIAL: NCT04174963
Title: An Electronic Intervention to Reduce Cannabis Among Young Adults in Psychiatric Care
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Based on Initial findings and input from other researchers in the field, the investigators and sponsor decided to end this study and begin work on an updated version of this research.
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Principal Investigator, Laura Whiteley, Assistant Professor, Rhode Island Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1445964
Record Dates: First submitted 2019-11-04; First posted 2019-11-22 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Cannabis Use; Psychiatric Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- eToke + TPsy (Experimental): All participants will receive the intervention (eToke+TPsy). The intervention consists of eToke (a brief computerized intervention that uses motivational enhancement therapy to improve readiness to decrease cannabis use and increase motivation to engage in substance use treatment) AND 6-8 interactive text messages regarding cannabis use reduction over 4 weeks . Text messages will contain written content, and queries, as well as links to publicly available websites and YouTube videos.
  Interventions: Behavioral: eToke + TPsy

INTERVENTIONS:
Behavioral: eToke + TPsy — Combination of brief computerized intervention (eToke) with Information-Motivation-Behavior based text messages tailored to young adults in psychiatric treatment

SUMMARY:
Cannabis use disorders are common among young adults in psychiatric treatment. Unfortunately, cannabis use can result in deleterious consequences for those in treatment, including developing more severe psychopathology and poorer treatment outcomes. Brief, electronic interventions for cannabis use have been developed for young adults. An example of a frequently used brief electronic intervention for cannabis users is e-Toke. e-Toke can be completed on a computer, tablet or phone, and has been shown to improve motivation to engage in substance use treatment among college students. However, e-Toke is less useful in decreasing the actual frequency of cannabis use. Additionally, e-toke is not tailored to young adults in psychiatric treatment. In this study, the investigators will develop and test a text messaging intervention that can be easily added to the popular computerized intervention e-Toke. The research staff hope the intervention will improve motivation to decrease cannabis use, and decrease the frequency of cannabis use, among young adults in psychiatric outpatient treatment. The text messages will be developed by, and tailored to, young adults in psychiatric treatment and texts will address motivations and barriers to reducing cannabis use in the context of psychiatric disorders. If the text message intervention is found to be an effective addition to e-Toke, this approach can be tested in a larger study, and then disseminated to other young adults in psychiatric treatment.

DETAILED DESCRIPTION:
Young adults 18-28 years old have the highest prevalence rates of cannabis use. Unfortunately, the biological consequences of cannabis use are more severe compared to older adults. These specific biological consequences are due to the negative effect cannabis use has on neurological maturation permanently impacting motivation, impulsivity, and future addictive behavior. The neurological effects of cannabis use are most disruptive to young adults living with psychiatric illness. In the Young Adult Behavioral Health Program at Rhode Island Hospital, 68% of patient's ages 18-28 who are in treatment for psychiatric disorders have used cannabis, and of those that have used 24% use cannabis daily or weekly. These high rates of cannabis use result in deleterious consequences, including developing more severe psychopathology, increased rates of psychosis, impairments in educational achievement and occupational obtainment, poorer treatment outcomes, poorer adherence to treatment, and increased treatment costs. Motivational Enhancement Therapy (MET) is an efficacious strategy for improving readiness to decrease cannabis use and increase motivation to engage in substance use treatment. The MET program entitled eToke (also known as E-Check-Up to Go), is a popular, frequently used, and previously investigated brief computerized intervention with efficacy in improving readiness for change among college students. In this study, the investigators propose to develop a text messaging intervention that will accompany eToke and will be tailored to young adults with psychiatric illness with cannabis use disorders. This intervention will be called e-Toke+TPsy. The text messages used in this intervention will contain information about the deleterious consequences of cannabis use, motivational material about the specific risks of cannabis use for young adults in psychiatric treatment. Texts will also contain behavioral skill building exercises to help reduce the frequency of cannabis use. The material for the text messages will be developed with input from young adults receiving psychiatric care at the Young Adult Behavioral Health Program. Text messages will also be informed by the Information, Motivation, and Behavioral Skills Theory of learning (IMB Theory).

ELIGIBILITY:
Inclusion Criteria:

* 18 - 28 years of age
* Report using cannabis 2 or more times per week
* English speaking
* Have a telephone that can receive text-messages
* Receive psychiatric treatment in the Young Adult Behavioral Health Program or Partial Program at Rhode Island Hospital.
* Be at high risk for psychosis according to mental health guidelines

Exclusion Criteria:

* Psychiatric symptoms severe enough to preclude meaningful consent or participation, as determined by the treatment psychiatrist and research team
* Current clinical diagnosis of mental retardation or pervasive developmental disorder

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
Change in Self-reported Frequency of Cannabis Use | Assessed at weeks 2, 4, 5, 6, 7, 8, 9, 10, and 11
  This self-report will be obtained using an abbreviated version of the Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST) nine times throughout the duration of the study. The abbreviated ASSIST will be administered at weeks 2, 4, 5, 6, 7, 8, 9, 10, and 11 of the study.
Change in Self-reported Motivation to Reduce Cannabis Use (SOCRATES) | Assessed at baseline and 12 weeks
  Motivation to change substance use will be assessed using the Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES) adapted for cannabis use (19-item questionnaires that assess recognition, ambivalence, and taking steps). Change will be assessed from baseline to 12-weeks follow-up.
Change in Self-reported Motivation to Reduce Cannabis Use (Readiness Ruler) | Assessed at baseline and 12 weeks
  Motivation to change substance use will be assessed using the Readiness Ruler (rates degree of readiness to cut down ranging from 1 to 10 for twelve different substance categories). Change will be assessed from baseline to 12-weeks follow-up.
Change in Self-reported Motivation to Reduce Cannabis Use (DBI) | Assessed at baseline and 12 weeks
  Motivation to change substance use will be assessed using the Decisional Balance Inventory (16-item measure of the pros and cons of substance use). Change will be assessed from baseline to 12-weeks follow-up.

SECONDARY OUTCOMES:
Change in Self-reported Psychiatric Symptoms | Assessed at baseline and 12 weeks
  Mental health issues will be assessed by the Brief Symptom Inventory (BSI-18), which yields primary symptom scales and global indices and has norms for adolescents and adults. The reliability, validity, and utility of the BSI instrument have been tested in more than 400 research studies. Internal consistency for the sub-scales (dimensions) range from .71 to .85. Each item will be reported on a scale of 0 to 4, with higher scores indicating greater mental health symptoms. Change will be assessed from baseline to 12-weeks follow-up.
Change in Self-reported Self-efficacy to Reduce Cannabis Use (SCQ-8) | Assessed at baseline and 12 weeks
  Self-efficacy will be assessed with the Situational Confidence Questionnaire (SCQ-8), an 8-item measure that assesses an individual's confidence in being able to resist the urge to use a given substance across different situations. The SCQ has been demonstrated reliable and valid. Each item is reported on a scale of 0 to 100, with higher scores indicating greater self-efficacy to resist using cannabis. Change will be assessed from baseline to 12-weeks follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Whiteley, MD, Principal Investigator — Rhode Island Hospital; Larry Brown, MD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Background] Elliott JC, Carey KB. Correcting exaggerated marijuana use norms among college abstainers: a preliminary test of a preventive intervention. J Stud Alcohol Drugs. 2012 Nov;73(6):976-80. doi: 10.15288/jsad.2012.73.976. PMID 23036216
- [Background] Miller WR, Tonigan JS. Assessing drinkers' motivation for change: The Stages of Change Readiness and Treatment Eagerness Scale (SOCRATES). Psychology of Addictive Behaviors 10(20): 81-89, 1996.
- [Background] Migneault JP, Pallonen UE, Velicer WF. Decisional balance and stage of change for adolescent drinking. Addict Behav. 1997 May-Jun;22(3):339-51. doi: 10.1016/s0306-4603(96)00252-3. PMID 9183504
- [Background] Derogatis LR, Melisaratos N. The Brief Symptom Inventory: an introductory report. Psychol Med. 1983 Aug;13(3):595-605. PMID 6622612
- [Background] Kirisci L, Moss HB, Tarter RE. Psychometric evaluation of the Situational Confidence Questionnaire in adolescents: fitting a graded item response model. Addict Behav. 1996 May-Jun;21(3):303-17. doi: 10.1016/0306-4603(95)00060-7. PMID 8883482
- [Background] WHO ASSIST Working Group. The Alcohol, Smoking and Substance Involvement Screening Test (ASSIST): development, reliability and feasibility. Addiction. 2002 Sep;97(9):1183-94. doi: 10.1046/j.1360-0443.2002.00185.x. PMID 12199834